CLINICAL TRIAL: NCT05826379
Title: Mechanisms of Adherence to Light Intensity Physical Activity to Prevent Alzheimer's Disease and Related Dementias (ADRD)
Brief Title: Daily Goal Setting to Increase Everyday Physical Activity and Promote Cognitive Health in Midlife
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jonathan Hakun, Assistant Professor of Neurology, Psychology, & Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY00022087; R61AG078084 (NIH)
Record Dates: First submitted 2023-03-15; First posted 2023-04-24 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Physical Inactivity; Walking; Cognitive Health; Self-regulation; Overweight and Obesity
MeSH Terms: conditions — Sedentary Behavior; Self-Control; Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Participants receive the adaptive daily step goal mHealth intervention
  Interventions: Behavioral: Adaptive Daily Goal Setting
- Treatment (Experimental): Participants receive the adaptive daily step goal mHealth intervention plus interim goal setting prompts each day
  Interventions: Behavioral: Adaptive Daily Goal Setting; Behavioral: Interim Goal Prompt

INTERVENTIONS:
Behavioral: Adaptive Daily Goal Setting — Daily step goals displayed by the study application
Behavioral: Interim Goal Prompt — Short-term step goals
  Arms: Treatment

SUMMARY:
The purpose of this study is to determine whether interaction with an adaptive Fitbit-based goal setting application can increase levels of everyday light intensity physical activity in middle-aged adults.

DETAILED DESCRIPTION:
The study is designed to examine the efficacy of a Fitbit-based, goal setting, mHealth intervention to increase light intensity physical activity. The study design is a 2-arm randomized controlled trial. Both groups will receive the underlying goal-setting intervention (adaptive daily step goals). The study involves 3 phases: a run-in ("calibration") phase, the intervention ("training") phase, and follow-up (1- and 12-months post-intervention).

To support goal maintenance our team has developed a Fitbit application designed to operate on the Fitbit Versa series watch as a 'clockface'. The application will first calibrate participants' average level of physical activity by recording daily step counts for a period of 14 days (calibration phase). After this period (and following a health education session) the application will begin delivering the underlying intervention to both treatment and control groups for a period of 1 month. The intervention is composed of daily step goals presented via the Fitbit clockface. Each day the application will suggest a daily step goal. The algorithm used to make these suggestions relies on the participant's own activity during the calibration period and is updated each day in study, ensuring all proposed step goals are within their existing repertoire. Follow-up assessments will be completed at 1- and 12-monts post-intervention.

Outcomes and moderators will be measured via activity monitors (the Fitbit application and activPals), surveys, and ecological momentary assessments (self-ratings and performance-based ambulatory cognitive assessments) conducted via the Mobile Monitoring of Cognitive Change ("M2C2") platform.

Some of the details of the intervention, algorithm, experimental manipulations, and outcomes have been omitted to preserve the scientific integrity of the study. These details will be added after the study is closed.

ELIGIBILITY:
Inclusion Criteria*:

* Between 30 and 70 years of age
* BMI ≥ 25

Exclusion Criteria*:

* Clinical diagnosis of ADRD or other neurodegenerative disease
* Health condition contraindicated for increased physical activity
* Medical conditions or medications that would prohibit participation in an exercise test (e.g., decompensated heart failure, severe aortic stenosis, uncontrolled arrhythmia, and acute coronary syndromes)
* Limitations in use of a smart phone (e.g., issues with manual dexterity or visual impairment)
* Inability to walk unassisted
* BMI > 50
* Plan to have surgery or other procedure over the next 12 months that could affect mobility or light intensity physical activity maintenance
* Concurrent participation in a weight loss, physical activity, or cognitive training trial
* Failure to comply with Run-in Period activity monitoring (<70% valid wear days for the Fitbit and activPal)
* Anyone who will not discontinue the use of their own personal smartwatch during the training period.
* Anyone who scores below 19 on the MoCA-B would not be randomized after the Run-in Calibration Period.

Note: The eligibility criteria are deliberately incomplete to preserve the scientific integrity of the study. These details will be added after study closure.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Short-term adherence | 1-month follow-up
  Average of 14-day step count totals collected via ActivPal monitors
Long-term adherence | 12-month follow-up
  Average of 14-day step count totals collected via ActivPal monitors

SECONDARY OUTCOMES:
Self-Monitoring Behavior | Daily during intervention period
  Number of times participant checks their step count progress per day
Change in Cognitive Health (Processing Speed) | Change in mean performance between the 2-week calibration phase and 12-month follow-up
  Change in performance on ambulatory cognitive assessments of processing speed (response time during the "Symbol Search" task). This task is administered twice daily (2 "sessions" per day) throughout the 2-week, baseline "calibration phase" and twice daily throughout the 2-week, 12-month follow-up phase. The outcome to be modeled is median response time to trials administered during each session. Aggregation of data collected over these 2-week data collection periods will be model-based (in other words, all 'session' data will be modeled nested within phase, within persons).
Change in Cognitive Health (Working Memory Binding) | Change in mean performance between the 2-week calibration phase and 12-month follow-up
  Change in performance on ambulatory cognitive assessments of working memory binding (corrected recognition rate during the "Color Shapes" task). This task is administered twice daily (2 "sessions" per day) throughout the 2-week, baseline "calibration phase" and twice daily throughout the 2-week, 12-month follow-up phase. The outcome to be modeled is corrected recognition rate (hit rate minus false alarm rate) for trials administered during each session. Aggregation of data collected over these 2-week data collection periods will be model-based (in other words, all 'session' data will be modeled nested within phase, within persons).
Change in Self-Efficacy for light intensity physical activity | Change between pre-enrollment baseline survey and end of training phase (an average of 2 months)
  Self-efficacy for exercise scale (adapted to light intensity physical activity; range 0-90 points; higher scores reflect better outcomes)
Executive Control (Working Memory Capacity) | Twice daily during the final 2 weeks of the training phase
  Performance on ambulatory cognitive assessments of working memory capacity (span score during the "Rotation Span" task). This task is administered twice daily (2 "sessions" per day) during the last 2 weeks of the "training phase". The outcome to be modeled is the total recalled arrows across the 3 trials assessed during each session. Data will not be aggregated, but instead modeled as a time-varying covariate.
Executive Control (Inhibitory Control) | Twice daily during the final 2 weeks of the training phase
  Performance on ambulatory cognitive assessments of inhibitory control (commission errors during the "Go/NoGo" task). This task is administered twice daily (2 "sessions" per day) during the last 2 weeks of the "training phase". The outcome to be modeled is the total commission errors across the trials assessed during each session. Data will not be aggregated, but instead modeled as a time-varying covariate.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan G Hakun, PhD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States